CLINICAL TRIAL: NCT06608446
Title: Effects of a Telerehabilitation Intervention in the Management of Complications After Breast Cancer Surgery: Randomized Controlled Trial
Brief Title: Effects of a Telerehabilitation Intervention in the Management of Complications After Breast Cancer Surgery
Acronym: LINFO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.032
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Telerehabilitation; Standard of Care

STUDY DESIGN:
Intervention Model Description: Non-profit blinded randomized controlled interventional single-center pilot study.
Who Masked: Outcomes Assessor
Masking Description: the evaluators do not know the treatment group of the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation (Experimental): In the days following surgery, intervention group will receive a structured rehabilitation session by a physiotherapist. In this session, two booklets will be provided to the patients, with the aim of informing and educating, regarding the most frequent complications after breast cancer surgery and how to avoid their possible onset through the demonstration of exercises to be carried out at home, self-massage techniques of the scar, behaviors and lifestyle to be adopted immediately after surgery.
  This group will carry out, starting from 10 days post-surgery, a home tele-rehabilitation intervention from Monday to Friday via the TeleHab device (Vald Performance) until 2 months after surgery.
  Exercises for ROM recovery and strength recovery will be carried out three days a week and only exercises for ROM recovery will be carried out two days a week.
  Interventions: Other: Telerehabilitation
- Standard care (Active Comparator): Standard care consists of the usual treatment according to current clinical practice, no structured physiotherapeutic interventions will be carried out which generally consists of the delivery of two booklets, with the aim of informing and educating, regarding the most frequent complications after breast cancer surgery and how to avoid its possible onset through the demonstration of exercises to be carried out at home, self-massage techniques for the scar, behaviors and lifestyle to be adopted immediately after surgery.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Telerehabilitation — The telerehabilitation intervention will begin from 10 days post-surgery, the operation will be carried out at home from Monday to Friday via the TeleHab device (Vald Performance) up to 2 months after the surgery.
  Exercises for ROM recovery and strength recovery will be carried out three days a week and only exercises for ROM recovery will be carried out two days a week. The progression of the exercises will be carried out taking into account the pain and fatigue recorded by the patient at the end of each exercise session.
  Arms: Telerehabilitation
Other: Standard Care — Standard care intervention follow the usual treatment according to current clinical practice, no structured physiotherapeutic interventions will be carried out. It consists of the delivery of two booklets, with the aim of informing and educating, regarding the most frequent complications after breast cancer surgery and how to avoid its possible onset through the demonstration of exercises to be carried out at home, self-massage techniques for the scar, behaviors and lifestyle to be adopted immediately after surgery.
  Arms: Standard care

SUMMARY:
The most common complaints after breast surgery are postoperative pain reported in up to 68% of patients, musculoskeletal problems in the shoulder and functional limitations in up to 59% of patients after mastectomy and quadrantectomy, reduction in range of motion ( ROM) in 24-53% and strength deficit.

The study aims to verify the effectiveness of a telerehabilitation treatment in terms of prevention of possible complications following breast cancer surgery.

Primary objective: to examine whether the group of patients undergoing rehabilitation surgery in the immediate post-operative period shows a reduction in the onset of complications compared to the group of patients who followed standard procedures.

Secondary objective: to study any preoperative prognostic factors for the onset of complications, to study the effectiveness of the rehabilitation treatment in terms of reduction of painful symptoms, improvement of joint ROM, muscle strength and perceived quality of life.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women worldwide. Advances in early detection and improved treatment of breast cancer have led to increased survival after diagnosis, resulting in many more women living with the consequences of cancer treatment.

Breast cancer surgeries and treatments can cause arm morbidity that can progress beyond 2.5 years.

The most common complaints after breast surgery are postoperative pain reported in up to 68% of patients, musculoskeletal problems in the shoulder and functional limitations in up to 59% of patients after mastectomy and quadrantectomy, reduction in range of motion ( ROM) in 24-53% and strength deficit.

Other complications include postoperative axillary web syndrome (AWS), which can cause pain and movement limitations; lymphedema reported with a prevalence of 6-52% especially after axillary lymph node dissection (ALND); kinematic alterations that may promote future development of rotator cuff disease; scapulohumeral dyskinesia, proprioception deficit, postural alterations and reduced quality of life.

There is scientific evidence in the literature to suggest that early postoperative exercise is safe and can improve shoulder function; however, uncertainty remains about the optimal content, timing, and cost-effectiveness of exercise interventions.

The study aims to verify the effectiveness of a rehabilitation treatment in terms of prevention of possible complications following breast cancer surgery.

Primary objective: to examine whether the group of patients undergoing rehabilitation surgery in the immediate post-operative period shows a reduction in the onset of complications compared to the group of patients who followed standard procedures.

Secondary objective: to study any preoperative prognostic factors for the onset of complications, to study the effectiveness of the rehabilitation treatment in terms of reduction of painful symptoms, improvement of joint ROM, muscle strength and perceived quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer
* Having undergone quadrantectomy or mastectomy surgery
* Age > 18 years
* Signature of informed consent

Exclusion Criteria:

* Neurological deficits with sensorimotor impairment of the upper limb
* Cognitive deficits that prevent the completion of questionnaires (MMSE>24)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Complications | 7-10 days after surgery
  Number of complications (i.e. axyllary web syndrome; lymphedema)
Complications | 2 months after surgery
  Number of complications (i.e. axyllary web syndrome; lymphedema)
Complications | 6 months after surgery
  Number of complications (i.e. axyllary web syndrome; lymphedema)

SECONDARY OUTCOMES:
Upper limb pain | before surgery
  Pain assessed through the numeric pain rating scale (0-10)
Upper limb pain | 7-10 days after surgery
  Pain assessed through the numeric pain rating scale (0-10)
Upper limb pain | 2 months after surgery
  Pain assessed through the numeric pain rating scale (0-10)
Upper limb pain | 6 months after surgery
  Pain assessed through the numeric pain rating scale (0-10)
Neck Disability | before surgery
  Neck related disability assessed through the questionnaire Neck Disabiltiy Index Value range (0% min disability - 100% max disability)
Neck Disability | 7-10 days after surgery
  Neck related disability assessed through the questionnaire Neck Disability Index Value range (0% min disability - 100% max disability)
Neck Disability | 2 months after surgery
  Neck related disability assessed through the questionnaire Neck Disability Index Value range (0% min disability - 100% max disability)
Neck Disability | 6 months after surgery
  Neck related disability assessed through the questionnaire Neck Disability Index Value range (0% min disability - 100% max disability)
Upperlimb Disability | before surgery
  Upperlimb related disability assessed through the questionnaire Disability of the arm, shoulder and hand (DASH) Value range (0% min disability - 100% max disability)
Upperlimb Disability | 7-10 days after surgery
  Upperlimb related disability assessed through the questionnaire Disability of the arm, shoulder and hand (DASH) Value range (0% min disability - 100% max disability)
Upperlimb Disability | 2 months after surgery
  Upperlimb related disability assessed through the questionnaire Disability of the arm, shoulder and hand (DASH) Value range (0% min disability - 100% max disability)
Upperlimb Disability | 6 months after surgery
  Upperlimb related disability assessed through the questionnaire Disability of the arm, shoulder and hand (DASH) Value range (0% min disability - 100% max disability)
Self-reported Quality of life | before surgery
  Impact on quality of life assessed through the questionnaire Short Form-36 Health Survey Value range (0 min QoL- 100 max QoL)
Self-reported Quality of life | 7-10 days after surgery
  Impact on quality of life assessed through the questionnaire Short Form-36 Health Survey Value range (0 min QoL- 100 max QoL)
Self-reported Quality of life | 2 months after surgery
  Impact on quality of life assessed through the questionnaire Short Form-36 Health Survey Value range (0 min QoL- 100 max QoL)
Self-reported Quality of life | 6 months after surgery
  Impact on quality of life assessed through the questionnaire Short Form-36 Health Survey Value range (0 min QoL- 100 max QoL)
Joint range of motion | before surgery
  upper limb and cervical range of motion assessed through digital goniometer
Joint range of motion | 7-10 days after surgery
  upper limb and cervical range of motion assessed through digital goniometer
Joint range of motion | 2 months after surgery
  upper limb and cervical range of motion assessed through digital goniometer
Joint range of motion | 6 months after surgery
  upper limb and cervical range of motion assessed through digital goniometer
Muscle strength | before surgery
  shoulder and neck muscle strength assessed through handheld dynamometer
Muscle strength | 7-10 days after surgery
  shoulder and neck muscle strength assessed through handheld dynamometer
Muscle strength | 2 months after surgery
  shoulder and neck muscle strength assessed through handheld dynamometer
Muscle strength | 6 months after surgery
  shoulder and neck muscle strength assessed through handheld dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No